CLINICAL TRIAL: NCT03938831
Title: Effect of Dexmedetomidine in Postoperative Delirium in Hip Surgery
Brief Title: Dexmedetomidine and Delirium in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Il Ok Lee, professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K2019-03 58-003
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Delirium, Dexmedetomidine, Postoperative PCA
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: randomized control
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Experimental): dexmedetomidine mixture with fentanyl-based PCA infusion for 2 days
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl-based PCA infusion
- control group (Placebo Comparator): Fentanyl-based PCA infusion for 2 days
  Interventions: Drug: Fentanyl-based PCA infusion

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine 0.5 micg/kg/hr infusion during operation and followed by 0.2 mic/kg/hr with fentanyl-based PCA mixture for 2 days
  Arms: dexmedetomidine group
Drug: Fentanyl-based PCA infusion — Fentanyl-based PCA infusion

SUMMARY:
Investigators investigates the effect of perioperative dexmedetomidine 0.5 ug/kg/hr followed by a postoperative continuous infusion fentanyl-based PCA(Patient-Controlled Analgesia) drug mixed with dexmedetomidine 0.2ug/kg/hr for two days on reducing postoperative delirium and postoperative rescue analgesics in elderly patients who undergo hip surgery. The other half of patients received fentanyl-based PCA only.

DETAILED DESCRIPTION:
Elderly patients are susceptible to postoperative delirium. Delirium occurs in 10~60% and is associated with longer hospital stays, increased costs, and morbidity. Postoperative delirium usually occurs 2~3 days after surgery. Intraoperative infusion of dexmedetomidine lacks preventing postoperative delirium in elderly noncardiac major surgery.

We hypothesized postoperative dexmedetomidine for two days as a mixture drug of fentanyl-based PCA could reduce the incidence of postoperative delirium. We compared this effect with other control group who received fentanyl-based PCA only.

We also investigate EEG patterns of patients during emergence and compared the EEG patterns who developed delirium postoperatively in PACU(Postanesthesia care unit) or general ward. Dexmedetomidine has analgesic effect. We expected postoperative dexmedetomidine has benefits of opioid sparing effects.

ELIGIBILITY:
Inclusion Criteria: over 65 yrs old elderly patient who undergo elective hip surgery and ASA(The American Society of Anesthesiologists) physical status I-III

Exclusion Criteria:

history of dementia, drug abuser, hypersensitivity to dexmedetomidine, fentanyl, propofol, disable to speech, reject the clinical study, hemodynamic instability during surgery, an illiterate, pregnancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-08-28 (Estimated)

PRIMARY OUTCOMES:
delirium | 2 days
  reduction of incidence of delirium

CONTACTS AND LOCATIONS:
Overall Officials: Il-Ok Lee, professor, Study Chair — Korea University Guro Hospital
Locations (1):
- KoreaUniversity Guro Hospital, Seoul, Guro-ku, South Korea